CLINICAL TRIAL: NCT03492255
Title: CYCLONES - CYClophosphamide LOw Dose and No Extra Steroid
Acronym: CYCLONES
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Significative difference between percentage of renal response (primary outcome) between the two study arms.
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CYCLONES
Record Dates: First submitted 2018-03-16; First posted 2018-04-10 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-04

CONDITIONS: Systemic Lupus Erythematosus (SLE)
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Cyclophosphamide; Methylprednisolone; Prednisone; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Eurolupus: Cyclophosphamide + Methylprednisolone + oral GC (Active Comparator): The EUROLUPUS group will receive Cyclophosphamide (6 doses of 500 mg / fortnightly) + 3 doses of Methylprednisolone (750 mg) initial + oral glucocorticoid (GC) (prednisone) ≤ 30 mg/day with a gradual reduction of 5 mg/month (EUROLUPUS). From the 3rd month, the group will receive oral mycophenolate mofetil (MMF) (2-3 g) until 6 months with gradual reduction of GC from 5 mg/month until the minimum dose of 5 mg/month.
  Interventions: Drug: Cyclophosphamide; Drug: Methylprednisolone; Drug: Prednisone; Drug: Mycophenolate Mofetil
- Cyclones Group: Cyclophosphamide+Methylprednisolone no oral GC (Experimental): CYCLONES Group will receive for 3 months Cyclophosphamide (6 doses of 500mg / fortnightly) + Methylprednisolone [500 mg (day 0 and day 15), 250 mg (day 30 and day 45) and 125 mg (day 60 and day 75)] without oral glucocorticoid (GC). From the third month, the group will receive only oral MMF (2-3 g) until the 6th month. Patients using GC ≤ 20 mg/day may enter the protocol with immediate reduction to 15 mg/day with a reduction of 5mg/month until complete withdrawal.
  Interventions: Drug: Cyclophosphamide; Drug: Methylprednisolone; Drug: Mycophenolate Mofetil

INTERVENTIONS:
Drug: Cyclophosphamide — Patients in both EUROLUPUS group and CYCLONES Group will receive for 3 months Cyclophosphamide (6 doses of 500mg/biweekly)
Drug: Methylprednisolone — Patients in EUROLUPUS group will receive Methylprednisolone [750 mg for three consecutive days).
  Patients in CYCLONES Group will receive Methylprednisolone [500 mg (day 0 and day 15), 250 mg (day 30 and day 45) and 125 mg (day 60 and day 75).
Drug: Prednisone — Patients in EUROLUPUS group will receive oral prednisone ≤ 30 mg/day with a reduction of 5mg/month until complete withdrawal.
  Arms: Eurolupus: Cyclophosphamide + Methylprednisolone + oral GC
Drug: Mycophenolate Mofetil — From the third month of protocol, patients in both EUROLUPUS group and CYCLONES Group will receive mycophenolate mofetil (2-3 g/day) until the sixth month of study.

SUMMARY:
Glucocorticoids (GC) use has increased survival of patients with systemic lupus erythematosus (SLE), particularly in cases of nephritis and a more significant improvement to 80% with the introduction of therapy combined with immunosuppressants. This therapeutic scheme, however, results in a very high incidence of irreversible damage that is associated in more than 70% of the cases to GC use and in a smaller proportion to the use of high dose cyclophosphamide.

CYCLONES is a Controlled Randomized Clinical Trial with the aim of evaluating the efficacy of a regimen for lupus nephritis treatment using only intravenous corticosteroid administration. This intravenous corticosteroid regimen has already been tested (with Rituximab instead of Cyclophosphamide) with high response rates for lupus nephritis and significant reduction of side effects.

After selection, patients will be randomized in two arms: 116 patients will receive Euro-Lupus nephritis regimen and other 116 will undergo treatment with CYCLONES regimen.

The primary endpoint is the partial response (protein/creatinine ratio < 3 with decrease at least of 50% of the initial value and increase of creatinine not higher than 15% of the initial value) or complete response (protein/creatinine ratio < 500 with decrease at least of 50% of the initial value and increase of creatinine not higher than 15% of the initial value in 6 months. Secondary outcome measures will be evaluated such as osteoporosis and bone metabolism parameters, ophthalmologic evaluation of the collateral effects related to glucocorticoids, lipid profile and therapy adherence.

DETAILED DESCRIPTION:
The use of glucocorticoids (GC) greatly increased the survival of patients with SLE, particularly in cases of nephritis and a more significant improvement to 80% with the introduction of therapy combined with immunosuppressants in the late 1960s. This therapeutic regimen, however, results in a very high incidence of irreversible damage to the patient that is associated in more than 70% of the cases to GC use and in a smaller proportion to the use of a high dose of cyclophosphamide. In the last years, some less toxic schemes have been proposed. The use of low-dose cyclophosphamide has been shown to have equal efficacy as high dose for the induction of remission of lupus nephritis with a fifteen-year follow-up.

Regarding GC, lower doses of methylprednisolone (MP) pulse have been shown to have similar efficacy and lower risk of infection. In addition, retrospective studies have found that high doses of oral GC during the induction period are associated with a higher incidence of side effects without a corresponding increase in efficacy . But it was only in 2013 that the first study was published that did not use oral GC in the treatment of lupus nephritis induction with excellent results.

In transplantation area, there are already several trials minimizing the use of GC proposing in the first days after transplantation the use the methylprednisolone (MP) IV pulse (day 1, 500mg, day 2, 250mg and day 3, 125mg) followed by oral GC for 4 days (60mg, 40mg, 30mg and 20mg). In this study, the same incidence of acute rejection occurred when compared to patients who were treated with oral GC for a prolonged period.

Regarding the route of administration of GC, it is important to emphasize that MP is three times more active through non-genomic pathway than through genomic pathway, which, in theory, results in a higher efficiency and lower collateral effect, when compared to the GC oral route that has similar potency through the two pathways. In addition, MP has a simpler and dose-proportional pharmacokinetics, whereas for oral prednisolone this kinetics is more complex and difficult to predict the dose required to achieve a specific concentration.

Therefore, the present study intends to evaluate the efficacy and adverse effects of cyclophosphamide (EUROLUPUS scheme) associated to usual GC dose compared with EUROLUPUS with no extra oral GC regimen.

The estimated number of patients was 116 patients for each arm (considering an error α = 0.05 and a power (1-β) of 80%).

In moderate flares, due to other systemic manifestations, the use of a maximum of 20mg / day of prednisone for 1 month and a progressive reduction of 5mg every 15 days until withdrawal is allowed. Other immunosuppressive, biological, intravenous immunoglobulin or plasmapheresis will be prohibited.

Regarding statistics, an Intention-To-Treat (ITT) analysis will be performed for the randomized patients, so that patients presenting side effects or low adherence to treatment will remain in the randomized group and will be evaluated at week 24.

The proportion of patients achieving complete and partial remission at week 24 will be compared by the chi-square test or the Fisher's exact test, as appropriate. The same statistical methodology will be applied to compare the number of events listed as secondary endpoints.

ELIGIBILITY:
Inclusion Criteria:

All the criteria below have to be completed:

1. Systemic lupus erythematosus (SLE) according to the American College of Rheumatology (ACR) classification criteria and/or SLICC: according to the thematic protocol (Petri M, et al., Arthritis Rheum, 2012);
2. Age ≥18 years;
3. Lupus Glomerulonephritis Class III, IV or V according to the International Society of Nephrology (ISN)/Renal Pathology Society (RPS) Classification confirmed on renal biopsy (according to the routine protocol of our outpatient clinic) performed up to 3 months to 1 year prior to selection;
4. Menopause or use contraception method;
5. Informed consent.

Exclusion Criteria:

1. Creatinine clearance < 40 ml/min calculated (Cockcroft & Gault);
2. Intolerance to medication;
3. Absolute neutrophil count < 1,000/mm3;
4. Pregnancy or breastfeeding;
5. Infection requiring hospitalization;
6. Patients who used Cyclophosphamide in the last 6 months or biological in the last year;
7. Thrombotic renal microangiopathy;
8. Chronic terminal renal disease and/or class VI biopsy;
9. Non-adhesion profile;
10. Need to use another therapeutic scheme;
11. GC dose in the last 3 months not greater than 20mg/day.

11.Central nervous system (CNS) disorders or hemolytic anemia and severe thrombocytopenia (< 50,000 platelets/mm3).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2018-04-12 (Actual); Primary Completion 2021-07-02 (Actual); Study Completion 2021-07-02 (Actual)

PRIMARY OUTCOMES:
Partial renal response | Six months
  The primary endpoint is partial renal response, a composition of: urinary protein/creatinine ratio < 3g/g with decrease of at least 50% of the initial value and increase of creatinine (mg/dL) not higher than 15% of the initial value
Complete renal response | Six months
  Complete renal response, according to a composition of: urinary protein/creatinine ratio < 0,5 (g/g) with decrease of at least 50% of the initial value and increase of creatinine (mg/dL) not higher than 15% of the initial value.

SECONDARY OUTCOMES:
Osteoporosis evaluation | 6 months
  Evaluation of osteoporosis by bone densitometry (DXA)
Bone structure evaluation | 6 months
  Evaluation of bone structure by high resolution peripheral quantitative computed tomography (HRpQCT)]
Glaucoma evaluation | 15 days, 30 days and 3 months
  Ophthalmologic evaluation for glaucoma secondary to glucocorticoids use
Cataract evaluation | 3 months
  Ophthalmologic evaluation for cataract secondary to glucocorticoids use
Change from baseline Total cholesterol at 6 months | Baseline and 6 months
  Lipid profile evaluation including total cholesterol in mg/dL
Change from baseline Low-density lipoprotein (LDL) at 6 months | Baseline and 6 months
  Lipid profile evaluation including Low-density lipoprotein (LDL) in mg/dL
Change from baseline High-density lipoprotein (HDL) at 6 months | Baseline and 6 months
  Lipid profile evaluation including High-density lipoprotein (HDL) in mg/dL
Change from baseline Triglycerides at 6 months | Baseline and 6 months
  Lipid profile evaluation including triglycerides in mg/dL
Change from baseline Anti-High-density lipoprotein (anti-HDL) at 6 months | Baseline and 6 months
  Lipid profile evaluation including anti-High-density lipoprotein (anti-HDL)
Therapy adherence by a self-report medication adherence measure (8-item Morisky Medication Adherence Scale) | Baseline
  Therapy adherence will be evaluated by a self-report medication adherence measure (8-item Morisky Medication Adherence Scale). A total score of all items are calculated with a sum score ranging from 0 to 8 for adherence. The scores will be trichotomized into the following 3 levels of adherence: high adherence (score 8), medium adherence (score 6 to <8), and low adherence (score <6).
Change from baseline Serum levels of prednisone using Area Under the Curve [AUC] at 30 days, 3 months and 6 months | Baseline, 30 days, 3 months and 6 months
  Serum levels of prednisone will be measured along the follow up using Area Under the Curve [AUC]

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - Rheumatology Division of Hospital das Clínicas da Faculdade de Medicina da Universidade de Sao Paulo, São Paulo, São Paulo
  - Hospital das Clinicas da Faculdade de Medicina da USP, São Paulo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Costenbader KH, Desai A, Alarcon GS, Hiraki LT, Shaykevich T, Brookhart MA, Massarotti E, Lu B, Solomon DH, Winkelmayer WC. Trends in the incidence, demographics, and outcomes of end-stage renal disease due to lupus nephritis in the US from 1995 to 2006. Arthritis Rheum. 2011 Jun;63(6):1681-8. doi: 10.1002/art.30293. PMID 21445962
- [Background] Gladman DD, Urowitz MB, Rahman P, Ibanez D, Tam LS. Accrual of organ damage over time in patients with systemic lupus erythematosus. J Rheumatol. 2003 Sep;30(9):1955-9. PMID 12966597
- [Background] Houssiau FA, Vasconcelos C, D'Cruz D, Sebastiani GD, Garrido Ed Ede R, Danieli MG, Abramovicz D, Blockmans D, Mathieu A, Direskeneli H, Galeazzi M, Gul A, Levy Y, Petera P, Popovic R, Petrovic R, Sinico RA, Cattaneo R, Font J, Depresseux G, Cosyns JP, Cervera R. Immunosuppressive therapy in lupus nephritis: the Euro-Lupus Nephritis Trial, a randomized trial of low-dose versus high-dose intravenous cyclophosphamide. Arthritis Rheum. 2002 Aug;46(8):2121-31. doi: 10.1002/art.10461. PMID 12209517
- [Background] Ruiz-Arruza I, Lozano J, Cabezas-Rodriguez I, Medina JA, Ugarte A, Erdozain JG, Ruiz-Irastorza G. Restrictive Use of Oral Glucocorticoids in Systemic Lupus Erythematosus and Prevention of Damage Without Worsening Long-Term Disease Control: An Observational Study. Arthritis Care Res (Hoboken). 2018 Apr;70(4):582-591. doi: 10.1002/acr.23322. Epub 2018 Mar 7. PMID 28704598
- [Background] Condon MB, Ashby D, Pepper RJ, Cook HT, Levy JB, Griffith M, Cairns TD, Lightstone L. Prospective observational single-centre cohort study to evaluate the effectiveness of treating lupus nephritis with rituximab and mycophenolate mofetil but no oral steroids. Ann Rheum Dis. 2013 Aug;72(8):1280-6. doi: 10.1136/annrheumdis-2012-202844. Epub 2013 Jun 5. PMID 23740227
- [Background] Petri M, Orbai AM, Alarcon GS, Gordon C, Merrill JT, Fortin PR, Bruce IN, Isenberg D, Wallace DJ, Nived O, Sturfelt G, Ramsey-Goldman R, Bae SC, Hanly JG, Sanchez-Guerrero J, Clarke A, Aranow C, Manzi S, Urowitz M, Gladman D, Kalunian K, Costner M, Werth VP, Zoma A, Bernatsky S, Ruiz-Irastorza G, Khamashta MA, Jacobsen S, Buyon JP, Maddison P, Dooley MA, van Vollenhoven RF, Ginzler E, Stoll T, Peschken C, Jorizzo JL, Callen JP, Lim SS, Fessler BJ, Inanc M, Kamen DL, Rahman A, Steinsson K, Franks AG Jr, Sigler L, Hameed S, Fang H, Pham N, Brey R, Weisman MH, McGwin G Jr, Magder LS. Derivation and validation of the Systemic Lupus International Collaborating Clinics classification criteria for systemic lupus erythematosus. Arthritis Rheum. 2012 Aug;64(8):2677-86. doi: 10.1002/art.34473. PMID 22553077
- [Background] Then Bergh F, Kumpfel T, Schumann E, Held U, Schwan M, Blazevic M, Wismuller A, Holsboer F, Yassouridis A, Uhr M, Weber F, Daumer M, Trenkwalder C, Auer DP. Monthly intravenous methylprednisolone in relapsing-remitting multiple sclerosis - reduction of enhancing lesions, T2 lesion volume and plasma prolactin concentrations. BMC Neurol. 2006 May 23;6:19. doi: 10.1186/1471-2377-6-19. PMID 16719908
- [Background] Ruiz-Irastorza G, Danza A, Khamashta M. Glucocorticoid use and abuse in SLE. Rheumatology (Oxford). 2012 Jul;51(7):1145-53. doi: 10.1093/rheumatology/ker410. Epub 2012 Jan 23. PMID 22271756
- [Background] Rohatagi S, Barth J, Mollmann H, Hochhaus G, Soldner A, Mollmann C, Derendorf H. Pharmacokinetics of methylprednisolone and prednisolone after single and multiple oral administration. J Clin Pharmacol. 1997 Oct;37(10):916-25. doi: 10.1002/j.1552-4604.1997.tb04266.x. PMID 9505983
- [Background] Levic Z, Micic D, Nikolic J, Stojisavljevic N, Sokic D, Jankovic S, Kendereski A, Mavra M. Short-term high dose steroid therapy does not affect the hypothalamic-pituitary-adrenal axis in relapsing multiple sclerosis patients. Clinical assessment by the insulin tolerance test. J Endocrinol Invest. 1996 Jan;19(1):30-4. doi: 10.1007/BF03347855. PMID 8851689
- [Background] Barkhof F, Tas MW, Frequin ST, Scheltens P, Hommes OR, Nauta JJ, Valk J. Limited duration of the effect of methylprednisolone on changes on MRI in multiple sclerosis. Neuroradiology. 1994 Jul;36(5):382-7. doi: 10.1007/BF00612124. PMID 7936181
- [Background] Contreras G, Pardo V, Leclercq B, Lenz O, Tozman E, O'Nan P, Roth D. Sequential therapies for proliferative lupus nephritis. N Engl J Med. 2004 Mar 4;350(10):971-80. doi: 10.1056/NEJMoa031855. PMID 14999109
- [Background] Petri M, Buyon J, Kim M. Classification and definition of major flares in SLE clinical trials. Lupus. 1999;8(8):685-91. doi: 10.1191/096120399680411281. PMID 10568907
- [Background] Gladman DD, Urowitz MB, Goldsmith CH, Fortin P, Ginzler E, Gordon C, Hanly JG, Isenberg DA, Kalunian K, Nived O, Petri M, Sanchez-Guerrero J, Snaith M, Sturfelt G. The reliability of the Systemic Lupus International Collaborating Clinics/American College of Rheumatology Damage Index in patients with systemic lupus erythematosus. Arthritis Rheum. 1997 May;40(5):809-13. doi: 10.1002/art.1780400506. PMID 9153540
- [Background] Appel GB, Contreras G, Dooley MA, Ginzler EM, Isenberg D, Jayne D, Li LS, Mysler E, Sanchez-Guerrero J, Solomons N, Wofsy D; Aspreva Lupus Management Study Group. Mycophenolate mofetil versus cyclophosphamide for induction treatment of lupus nephritis. J Am Soc Nephrol. 2009 May;20(5):1103-12. doi: 10.1681/ASN.2008101028. Epub 2009 Apr 15. PMID 19369404
- [Background] Vincenti F, Schena FP, Paraskevas S, Hauser IA, Walker RG, Grinyo J; FREEDOM Study Group. A randomized, multicenter study of steroid avoidance, early steroid withdrawal or standard steroid therapy in kidney transplant recipients. Am J Transplant. 2008 Feb;8(2):307-16. doi: 10.1111/j.1600-6143.2007.02057.x. PMID 18211506